CLINICAL TRIAL: NCT05571254
Title: The Management of Transient Loss of Consciousness (TLOC) and Suspected Syncope in European Emergency Departments: a Prospective Cohort Study
Brief Title: The Management of Transient Loss of Consciousness and Suspected Syncope in European Emergency Departments
Acronym: SEED
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC22033
Record Dates: First submitted 2022-09-26; First posted 2022-10-07 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-09

CONDITIONS: Syncope
Keywords: syncope; transient loss of consciousness; emergency department
MeSH Terms: conditions — Syncope; Emergencies | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — All patients will have a focussed Case Report Form completed collecting routine data describing the prevalence, clinical presentation, assessment, management and ESC risk category of patients, at the time or shortly after the patients ED attendance.

SUMMARY:
Prospective multi centre cohort study examining the clinical presentation, diagnostic tests, and management of adult Emergency Department (ED) patients presenting with Transient Loss of Consciousness (TLOC) either undifferentiated or thought to be of syncopal origin.

DETAILED DESCRIPTION:
Syncope is a common ED problem. The three underlying causes are reflex (simple faint), orthostatic hypotension (blood pressure fall on standing) and cardiac disease (structural heart disease or cardiac dysrhythmia). Diagnosis is difficult and is not apparent in ~50% of patients after assessment. For the first time, European Society of Cardiology (ESC) guidelines incorporating ED management of patients presenting with TLOC, either undifferentiated or thought to be of syncopal origin, have been produced.

However, very little is currently known about the use of diagnostic algorithms and management of this patient group in EDs across Europe. As a result, the application of guidelines and the management of TLOC by European Society of Emergency Medicine (EUSEM) members in different countries and hospitals, cannot yet be recommended for use in settings other than those where they have been successfully validated.

This study aims to describe the prevalence, clinical presentation, current assessment, management strategies and ESC risk categories of patients presenting with TLOC (undifferentiated or thought to be of syncopal origin) to the ED, and will provide data to help identify the gaps in our knowledge and practice, and areas where further research and development work is required to fully implement European Society of Cardiology (ESC) guidelines within European EDs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) assessed in the ED with TLOC thought to be of syncopal origin.

Exclusion Criteria:

* Inability to consent
* Patient in custody or prison
* Aged <18 years
* TLOC thought to be due to neurological seizure (e.g., epilepsy/alcohol or drug withdrawal) or trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years of age and older presenting to the ED over a two-week period with TLOC, either undifferentiated or thought to be of syncopal origin.
Sampling Method: Non-Probability Sample
Enrollment: 952 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Participant age | Admission
  Participant age
Participant gender | Admission
  Participant gender
Mode of arrival | Admission
  Mode of arrival
Referral source | Admission
  Referral source
Presence of any European Society of Cardiology (ESC) syncope high-risk history features | Admission
  Which European Society of Cardiology syncope high-risk history features are present
ESC high-risk 'past medical history' features | Admission
  Which European Society of Cardiology syncope high-risk 'past medical history' features are present
Other medical comorbidities | Admission
  Other medical comorbidities
Rockwood Clinical Frailty Scale score | Admission
  Rockwood Clinical Frailty Scale is a well validated score ranging from 1 (Very Fit) to 9 (Terminally Ill) with defined descriptions for each category.
ESC high risk 'physical examination' factors | Admission
  ESC high risk 'physical examination' factors
Blood pressure (BP) on admission | Admission
  First Blood pressure (BP) measure in the Emergency Department in mmHg
Pulse rate on admission | Admission
  First pulse rate measured in the Emergency Department in beats per minute
Lying/standing systolic BP difference on admission | Admission
  First lying/standing systolic BP difference measured in the Emergency Department in mmHg
Number of participants with abnormal Electrocardiogram (ECG) readings | Admission
  Number of participants with abnormal ECG readings
Troponin levels | Admission
  Troponin levels
D-dimer levels | Admission
  D-dimer levels
Copeptin levels | Admission
  Copeptin levels
Natriuretic peptides levels | Admission
  Natriuretic peptides levels
ED clinician diagnosis | Admission
  ED clinician diagnosis - descriptive
Patient destination | Admission
  Descriptive options: Admitted to Observation/Clinical Decision Unit/Same Day Emergency Care unit/hospital floor with telemetry monitoring/hospital floor with no telemetry monitoring. Discharged to outpatient follow up/family doctor/General Practitioner care/home with no follow up
Reason(s) for admission | Admission
  Reason(s) for admission
Whether driving and occupation advice given | Admission
  Whether driving and occupation advice given
Status at discharge from hospital | 30 days
  Status at discharge from hospital
Length of hospital stay in days | 30 days
  Length of hospital stay in days
Hospital discharge diagnosis | 30 days
  Hospital discharge diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Matt Reed, Study Chair — University of Edinburgh
Locations (57):
- Albania (5):
  - Regional Hospital Durres, Durrës
  - Regional Hospital Centre "Xh. Kongoli" Elbasan, Elbasan
  - Spitali "Petro Nako" Sarandra, Sarandë
  - Regional Hospital Shkoder, Shkodër
  - University Hospital Centre "Mother Theresa" Tirana, Tirana
- Austria (2):
  - Allgemeines Krankenhaus der Stadt Wien/ Universitätskliniken, Vienna
  - Klinik Donaustadt, Vienna
- Belgium (4):
  - AZ Sint Jan Brugge, Bruges
  - AZ Alma Eeklo, Eeklo
  - Ghent University Hospital, Ghent
  - Heilig Hartziekenhuis Lier, Lier
- Czechia (2):
  - University Hospital Hradec Králové, Králová
  - University Hospital Královské Vinohrady, Prague
- Denmark (5):
  - Regionshospitalet Gødstrup, Herning
  - Nordsjællands Hospital, Hillerød
  - Regionshospitalet Randers, Randers
  - Sjællands Universitetshospital, Roskilde
  - Regionshospitalet Midt, Vildbjerg
- Kanta-Häme Central Hospital, Helsinki, Finland
- France (5):
  - CHU Besançon, Besançon
  - CHU Caen, Caen
  - CHU Clermond-Ferrand, Clermont-Ferrand
  - Medipole, Lyon
  - CHU Tours, Tours
- Greece (3):
  - University General Hospital ATTIKON, Athens
  - General Hospital Venizeleio, Heraklion
  - AHEPA Univesrity General Hospital of Thessaloniki, Thessaloniki
- Semmelweis University Department of Emergency Medicine, Budapest, Hungary
- Italy (5):
  - ED Azienda Ospedaliera Universitaria di Bologna (Sant'Orsola Hospital), Bologna
  - ED Azienda Ospedaliera-universitaria di Catania (San Marco Hospital), Catania
  - ED Azienda USL Toscana Centro, Firenze (San Giovanni di Dio Hospital), Florence
  - Azienda Ospedaliera di Perugia (Santa Maria Della Misericordia Hospital), Perugia
  - ED Azienda Ospedaliera-Universitaria integrata (Borgo Trento Hospital), Verona
- Malta (2):
  - Mater Dei Hospital, Birkirkara
  - Gozo General Hospital, Victoria
- St. Olav's University Hospital, Trondheim, Norway
- Wroclaw University Hospital, Wroclaw, Poland
- Romania (2):
  - Cluj Napoca County Emergency Clinical Hospital, Cluj-Napoca
  - Saint Spiridon County Hospital, Iași
- Serbia (3):
  - Emergency Center Belgrade, Clinical Centre Belgade, Belgrade
  - Clinical Centre of Niš, Niš
  - Emergency Department Zaječar, Health Center Zaječar, Zaječar
- Spain (5):
  - Hospital Dr. Balmis, Alicante
  - Hospital clinic Barcelona, Barcelona
  - Hospital de Terrassa, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari de Vic, Barcelona
- Turkey (Türkiye) (5):
  - Gazi University Medical Faculty Department of Emergency Medicine, Ankara
  - Medical Science University Ankara Education and Research Hospital Department of Emergency Medicine, Ankara
  - Karamanoglu Mehmetbey University Karaman Education and Research Hospital Department of Emergency Medicine, Karaman
  - Necmettin Erbakan University Medical Faculty Department of Emergency Medicine, Konya
  - Medical Science University Sanliurfa Mehmet Akif Inan Education and Research Hospital Department of Emergency Medicine, Sanliurfa
- United Kingdom (5):
  - Royal Infirmary of Edinburgh, Edinburgh, Midlothian
  - University Hospital Coventry & Warwickshire, Coventry
  - Victoria Hospital, Kirkcaldy
  - St Johns Hospital, Livingston, Livingston
  - Royal Preston Hospital, Preston

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reed MJ, Karuranga S, Kearns D, Alawiye S, Clarke B, Mockel M, Karamercan M, Janssens K, Riesgo LG, Torrecilla FM, Golea A, Fernandez Cejas JA, Lupan-Muresan EM, Zaimi E, Nuernberger A, Rennet O, Skjaerbaek C, Polyzogopoulou E, Imecz J, Groff P, Camilleri R, Cimpoesu D, Jovic M, Miro O, Anderson R, Laribi S; SEED investigators. Management of syncope in the Emergency Department: a European prospective cohort study (SEED). Eur J Emerg Med. 2024 Apr 1;31(2):136-146. doi: 10.1097/MEJ.0000000000001101. Epub 2023 Nov 27. PMID 38015745